CLINICAL TRIAL: NCT00341679
Title: Studies of the Natural History and Pathogenesis of Autoimmune/Connective Tissue Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905200; 05-E-N200
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-07-08

CONDITIONS: Autoimmune/Connective Tissue Diseases; Idiopathic Inflammatory Myopathies; Polymyositis; Dermatomyositis
Keywords: Autoimmune Diseases; Polymyositis; Dermatomyositis; Idiopathic Inflammatory Myopathies; CONNECTIVE TISSUE DISEASES; Natural History; IIM
MeSH Terms: conditions — Connective Tissue Diseases; Myositis; Polymyositis; Dermatomyositis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family Members: Family members need to be blood relatives of the proband with the diagnosis of an autoimmune disease
- IIM Patient: Adult and pediatric patients with diagnosis of myositis or a related autoimmune or rheumatic disorder (by Bohan and Peter criteria, American College of Rheumatology, or other criteria).
- Normal volunteers: gender and race-matched to a subset of autoimmune subjects as controls. Should be without any autoimmune disease.

SUMMARY:
This study will define the major genetic risk and protective factors for idiopathic inflammatory myopathies (IIM), a group of immune disorders affecting connective tissues such as muscles. It will also identify new environmental risk factors for IIM and identify immune responses in myositis and related diseases. There are many forms of IIMs, and the causes of these diseases are unknown. However, scientists suspect that they result when people with some genetic factors that predispose them-that is, put them at greater risk-are exposed to certain environmental triggers. Some of those triggers include food, drugs, biologics (such as a vaccine to prevent disease), medical devices and occupational exposures.

Patients, including children under 18, who had a diagnosis of myositis, a related autoimmune disease, or a rheumatic disease, as well as their blood relatives, and control subjects who were in good health have already been recruited for this study.

The evaluation consisted of one outpatient visit to the patient's doctor, who will obtain a medical history and conduct a physician examination. Patients spent 20 to 30 minutes to answer written questions. There was a blood collection of about 6 tablespoons. If there was a major change in patients' medical conditions, they were asked to return for a second outpatient evaluation to determine whether any of the blood tests or antibodies, which show an immune response, had changed. Blood samples collected will be used only for laboratory research studies. The samples have been identified by a code, and all other identifying information have been removed.

During the study, researchers will explore possible environmental risk factors, including studies of infectious and non-infectious agents. They will analyze the blood for genetic markers and test for certain antibodies. Laboratory results will be evaluated as they relate to the signs, symptoms, and severity of patients' illnesses. That would help researchers to better understand patterns of the diseases and the outcomes for patients.

This study will not have a direct benefit for patients. However, results from the study can be made available to patients' doctors for use in appropriate care. Also, it is hoped that information gained can help other people in the future.

...

DETAILED DESCRIPTION:
Individuals who develop chronic harmful inflammation in association with self-reactive autoantibodies or T cells are said to have autoimmune diseases. The causes of these diseases are unknown but they are thought to occur in genetically susceptible individuals after exposure to selected environmental agents. There are many forms of these diseases, but we have been focusing on one of the rarest and most poorly-studied group of autoimmune disorders, known as the Idiopathic Inflammatory Myopathies (IIM). This heterogeneous group of diseases includes polymyositis, dermatomyositis and related disorders. This is a natural history protocol designed to continue our study of these diseases and begin the evaluation of related connective tissue disorders associated with environmental exposures. We plan to further delineate important groups of patients and familial cases, and obtain useful material for further investigations of the clinical presentations, etiology, pathogenesis, and immunologic abnormalities of autoimmune/connective tissue diseases. Clinical data and patient blood, urine and tissue specimens have been collected by referring physicians and sent to us. The blood samples have been separated into cells and plasma, frozen and then placed into cell and plasma banks. Often the diagnosis of an IIM can be confused with other illness (such as adult-onset dystrophies), and therefore, we have also included patients with other illnesses (who are referred with a preliminary diagnosis of an IIM or an unknown myopathy), including patients with other autoimmune diseases. In order to understand more fully the genetic risk factors for these diseases, family members of selected patients who have several blood relatives with autoimmune or connective tissue diseases will also be studied. In summary, this natural history protocol will attempt, through a series of hypothesis-testing and hypothesis-generating studies, to obtain new information regarding the clinical presentation, risk and protective factors, pathogeneses and prognostic features for myositis and related conditions.

ELIGIBILITY:
* Recruitment into the study is by invitation.

INCLUSION CRITERIA:

For the primary autoimmune and myositis study populations, children (less than 18 years of age) or adults (18 or more years of age) require a diagnosis of myositis or a related autoimmune or rheumatic disorder.

Family members need to be blood relatives of the proband with the diagnosis of an autoimmune disease.

Normal volunteers will be gender- and race-matched to a subset of autoimmune subjects as controls needed for specific studies.

Normal volunteers should be in good health, without a recognized systemic rheumatic disorder or other autoimmune disease, and should not be taking anti-inflammatory medicines, including nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.

For all subjects: ability of the subject or parents/legal guardians to provide informed consent to all aspects of the study after full protocol information is provided.

Patients enrolling in the MYOVISION national myositis patient registry were diagnosed with adult or juvenile DM, PM, IBM, or another form of myositis; resided within the United States or Canada at the time of diagnosis, and provided informed consent and completed the study questionnaires, either on paper or online. In the case of children <18 years of age, the parent or legal guardian provided informed consent and completed the study questionnaires.

EXCLUSION CRITERIA:

Exclusion criteria for all protocol subjects:

1. medical illness that in the judgment of the investigators does not allow safe blood draws or other clinical evaluations needed for study participation;
2. cognitive impairment;
3. inability to give informed assent or consent.

Exclusion criteria for normal volunteers:

Recognized systemic rheumatic disorder or other autoimmune disease, history of cancer or taking anti-inflammatory medicines, including nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids, severe trauma, infections or vaccinations within 8 weeks.

Exclusion criteria for patients in the MYOVISION national myositis patient registry were subjects with cognitive impairment and those unable to or unwilling to give informed consent,or failing to meet the inclusion criteria of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children (< 18 years of age) or adults (18 or more years of age) require a diagnosis of myositis or a related autoimmune or rheumatic disorder (by Bohan and Peter, American College of Rheumatology, or other criteria. Family members need to be blood relatives of the proband with the diagnosis of an autoimmune disease. Selected patients with other myopathies or with undefined illnesses who may have weakness, myalgias, or an elevated CK may be evaluated to establish a diagnosis. Normal volunteers will be gender- and race-matched to a subset of autoimmune subjects as controls needed for specific studies. Normal volunteers should be in good health, without a recognized systemic rheumatic disorder or other autoimmune disease, and should not be taking anti-inflammatory medicines, including non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2005-07-13 (Actual)

PRIMARY OUTCOMES:
Myositis Autoantibodies | at the time of enrollment visit
  Individuals who develop autoimmune diseases are associated with self-reactive autoantibodies. The clinical course of disease in IIM appears to be more closely related to the presence of certain myositis-specific autoantibodies
Human leukocyte antigen | at the time of enrollment visit
  The efforts to identify candidate genes will initially include polymorphic MHC and non-MHC immune response genes such as those for HLA,cytokines and chemokines with the strongest known associations with autoimmunity

SECONDARY OUTCOMES:
Environmental Exposures | ongoing
  Assessment of possible selected environmental risk factors will include studies of infectious and non-infectious agents by immunologic and other approaches. Birthdates, seasonal and geographic associations with disease onset, as well as unusual clustering in the frequencies of selected phenotypes or genotypes will also be studied.
Clinical Phenotyping of | ongoing
  The different phenotypes and immunologic abnormalities found in the clinicopathologic and immune response groups of the IIM suggest possible different pathogenesis and risk factors.
Pathogenesis of the Disease | ongoing
  to find possible different pathogenesis of multiple immune-mediated disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Rider, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institute of Environmental Health Sciences (NIEHS), 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study team is still deciding if they would like to share individual participant data

REFERENCES:
- [Background] Rider LG, Shah M, Mamyrova G, Huber AM, Rice MM, Targoff IN, Miller FW; Childhood Myositis Heterogeneity Collaborative Study Group. The myositis autoantibody phenotypes of the juvenile idiopathic inflammatory myopathies. Medicine (Baltimore). 2013 Jul;92(4):223-243. doi: 10.1097/MD.0b013e31829d08f9. PMID 23877355
- [Background] O'Hanlon TP, Carrick DM, Targoff IN, Arnett FC, Reveille JD, Carrington M, Gao X, Oddis CV, Morel PA, Malley JD, Malley K, Shamim EA, Rider LG, Chanock SJ, Foster CB, Bunch T, Blackshear PJ, Plotz PH, Love LA, Miller FW. Immunogenetic risk and protective factors for the idiopathic inflammatory myopathies: distinct HLA-A, -B, -Cw, -DRB1, and -DQA1 allelic profiles distinguish European American patients with different myositis autoantibodies. Medicine (Baltimore). 2006 Mar;85(2):111-127. doi: 10.1097/01.md.0000217525.82287.eb. PMID 16609350
- [Background] Miller FW, Chen W, O'Hanlon TP, Cooper RG, Vencovsky J, Rider LG, Danko K, Wedderburn LR, Lundberg IE, Pachman LM, Reed AM, Ytterberg SR, Padyukov L, Selva-O'Callaghan A, Radstake TR, Isenberg DA, Chinoy H, Ollier WE, Scheet P, Peng B, Lee A, Byun J, Lamb JA, Gregersen PK, Amos CI; Myositis Genetics Consortium. Genome-wide association study identifies HLA 8.1 ancestral haplotype alleles as major genetic risk factors for myositis phenotypes. Genes Immun. 2015 Oct;16(7):470-80. doi: 10.1038/gene.2015.28. Epub 2015 Aug 20. PMID 26291516